CLINICAL TRIAL: NCT04164914
Title: Intestinal Microbiota Adaptation to Prebiotic Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR(AG)420-2018
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Healthy
Keywords: intestinal gas; healthy subjects; microbiota; prebiotics
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Prebiotic administration
  Interventions: Dietary Supplement: Prebiotic

INTERVENTIONS:
Dietary Supplement: Prebiotic — Soluble prebiotic fiber (resistant dextrin 14 g/d x 4 weeks)

SUMMARY:
Non-absorbable, fermentable residues in the diet increase intestinal gas production and induce gas-related symptoms, such as flatulence, abdominal bloating and distention; however, prebiotics, which are also fermented by colonic bacteria, have been shown to improve this type of symptoms. The aim is to demonstrate whether a prebiotic induces adaptive changes in metabolic activity of gut microbiota and colonic biomass that explain its beneficial effect on gas-related symptoms.

Single-centre, single arm, open label, proof-of-concept study in healthy subjects. The study will consist of a pre-administration phase (2 wk), an administration phase (4 wk) and a post-administration phase (2 wk). A soluble prebiotic fiber (resistant dextrin 14 g/d) will be administered during the 4 wk administration phase. During 4 days immediately before, at the beginning and at the end of the administration phase and at the end of the post-administration phase participants will be put on a standard diet and the following outcomes will be measured: a) number of gas evacuations during daytime for 2 days by means of an event marker; b) volume of gas evacuated via a rectal tube during 4 hours after a test meal, by means of a barostat; c) microbiota composition by fecal analysis.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* gastrointestinal symptoms
* recent (3 months) antibiotic intake
* change in dietary habits 4 weeks before

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of daily anal gas evacuations | 28 days
  Change in the number of anal gas evacuations measured by an event marker from beginning of treatment to end of treatment

SECONDARY OUTCOMES:
Volume of anal gas evacuation | 28 days
  Change in the volume of anal gas evacuated for 4 hours after a probe meal from beginning of treatment to end of treatment
Microbiota composition by fecal analysis | 28 days
  Change from beginning of treatment to end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron Research Institut, Barcelona, Spain